CLINICAL TRIAL: NCT05739786
Title: Comparison of Efficacy of Liquid Nitrogen Versus Vitamin D3 in The Treatment of Cutaneous Warts
Brief Title: Comparisom of Liquid Nitrogen and Vitamin D3 in The Treatment of Cutaneous Warts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Sara Ilyas, principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CMHAtd-ETH-17-DERM-22
Record Dates: First submitted 2023-01-18; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Cutaneous Warts
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A liquid nitrogen (Active Comparator): liquid nitrogen In Group A patients were subjected to liquid nitrogen cryotherapy (-196 0C) for 3 sessions at every 3 weeks interval. Effectiveness in was ascertained in terms of > 50% reduction in wart size by an expert dermatologist on physical examination at the end of third session. Patients were followed for further 6 weeks after last session to look for any sort of recurrence and remission.
  Interventions: Drug: liq nitrogen
- Group B intralesional Vit D3 (Active Comparator): intralesional Vit D3 Group B were subjected to vitamin D3 (5mg/ml) for 3 sessions at every 3 weeks interval. Effectiveness was ascertained in terms of > 50% reduction in wart size by an expert dermatologist on physical examination at the end of third session. Patients were followed for further 6 weeks after last session to look for any sort of recurrence and remission.
  Interventions: Drug: intralesional vitamin D3

INTERVENTIONS:
Drug: liq nitrogen — In Group A patients were subjected to liquid nitrogen cryotherapy (-196 0C) for 3 sessions at every 3 weeks interval. Effectiveness in was ascertained in terms of > 50% reduction in wart size by an expert dermatologist on physical examination at the end of third session. Patients were followed for further 6 weeks after last session to look for any sort of recurrence and remission.
  Other Names: cryotherapy
  Arms: Group A liquid nitrogen
Drug: intralesional vitamin D3 — Group B were subjected to vitamin D3 (5mg/ml) for 3 sessions at every 3 weeks interval. Effectiveness was ascertained in terms of > 50% reduction in wart size by an expert dermatologist on physical examination at the end of third session. Patients were followed for further 6 weeks after last session to look for any sort of recurrence and remission.
  Arms: Group B intralesional Vit D3

SUMMARY:
A total of 60 female patients (30 patients in each group) with cutaneious warts diagnosed by a consultant dermatologist on physical examination were included in this study.

In Group A patients were subjected to liquid nitrogen cryotherapy (-196 0C) while patients in Group B were subjected to vitamin D3 (5mg/ml) for 3 sessions at every 3 weeks interval. Effectiveness in both groups was ascertained in terms of > 50% reduction in wart size by an expert dermatologist on physical examination at the end of third session. Patients were followed for further 6 weeks after last session to look for any sort of recurrence and remission.

ELIGIBILITY:
Inclusion Criteria:

* Patient of cutaneous warts presented in dermatology department.

Exclusion Criteria:

* Immunosuppressed patients
* chronic skin diseases like eczema or autoimmune disease
* diabetes mellitus
* cold sensitivity , skin allergies
* pregnancy, and lactation
* periungual warts

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness of liquid nitrogen and intralesional vitamin D3 in treatment of cutaneous warts | 9 weeks
  For 2nd Article: A total of 60 female patients (30 patients in each group) with cutaneous warts diagnosed by a consultant dermatologist on physical examination were included in this study.
  In Group A patients were subjected to liquid nitrogen cryotherapy (-196 0C) while patients in Group B were subjected to vitamin D3 (5mg/ml) for 3 sessions at every 3 weeks interval. Effectiveness in both groups was ascertained in terms of > 50% reduction in wart size by an expert dermatologist on physical examination at the end of third session. Patients were followed for further 6 weeks after last session to look for any sort of recurrence and remission.Total duration of therapy for each patient will be 9 weeks after "recurrence and remission"

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Ilyas, Abbottābād, Kpk, Pakistan